CLINICAL TRIAL: NCT05629078
Title: Vision and Balance Changes After Bilateral Implantation of Toric Versus Non-Toric Intraocular Lenses in Cataract Patients With Astigmatism
Brief Title: Vision and Balance Changes After Bilateral Implantation of Toric IOLs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: Carl Zeiss Meditec AG (Industry); Glasgow Caledonian University (Other); University of St Mark and St John Plymouth (Unknown); University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Phillip J Buckhurst, Professor, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 286913
Record Dates: First submitted 2021-03-04; First posted 2022-11-29 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cataract Bilateral; Astigmatism Bilateral
Keywords: toric intraocular lens; dynamic stability; balance; post-cataract surgery; fear of falling; visual function; quality of life
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: randomised control trial
Who Masked: Investigator
Masking Description: investigators will be blinded to which types of IOLs implanted to the cataract patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toric Intraocular lens (Active Comparator): Toric intraocular lens- AT TORBI® 709M, to be implanted bilaterally in the cataract surgery to correct astigmatism at the same time.
  Interventions: Device: Toric intraocular lens Zeiss AT TORBI
- Monofocal intraocular lens (Active Comparator): Standard monofocals IOLs- Zeiss CT ASPHINA 409/509M, to be implanted bilaterally in the standard NHS cataract surgery without correcting the astigmatism.
  Interventions: Device: Toric intraocular lens Zeiss AT TORBI

INTERVENTIONS:
Device: Toric intraocular lens Zeiss AT TORBI — Intraocular lenses are medical devices that are implanted in patients during cataract surgery. At Plymouth University NHS trust the standard lens is a monofocal non-Toric lens unless the patient has astigmatism greater than 4.00D. This study involves implantation of a toric lens in the intervention group where astigmatism is greater than 1.00D. The lens is called the toric IOLS- Zeiss AT TORBI, will be implanted bilaterally instead of standard monofocal IOLs- Zeiss CT ASPHINA, used in routine cataract surgery within NHS.
  Other Names: Monofocal non-toric intraocular lens Zeiss CT ASPHINA 409/509M

SUMMARY:
Cataracts are the major cause of blindness in the world. Cataract surgery, being the most performed surgery in the world today, provide correction by extracting the natural lens from its capsular bag and replaced by an artificial intraocular lens (IOL) implantation. In the UK, almost all patients undergoing cataract surgery by the NHS are given monofocal intraocular lenses (IOLs) which do not correct corneal astigmatic error. It is estimated that around 20% of the population has over 1.50DC of corneal astigmatism. Uncorrected astigmatism not only increase spectacle dependency and reduce quality of life post surgically, but it also adversely affects the overall economic costs. Specialised toric IOLs offer the opportunity to correct pre-existing corneal astigmatism. Previous work has shown a link between reduced vision and balance or mobility. Full correction of refractive error may have greater impact on lifestyle than previously thought.

DETAILED DESCRIPTION:
This is a single centre, parallel randomized controlled trial study comparing the dynamic stability and visual outcomes of cataract patient with astigmatism implanted with mono-focal Toric versus non-Toric IOLs.

140 cataracts patients with astigmatism awaiting cataract correction surgery at the Royal Eye infirmary of the University Hospitals of Plymouth NHS Trust will be recruited in this study over a two year period. The participants will be randomly assigned to be implanted with either Toric IOLs or standard non-Toric IOLs. Three additional study visits will be arranged for them. One visit before the cataract surgery, second visit at three to six months after the first eye cataract surgery and third visit at three to six months after the second eye cataract surgery. The primary assessment outcome is dynamic balance measured by movement sensors (accelerometer) during walk and turn, crossing over obstacle and stair walking. The secondary outcomes include eye tracking during movement activities, visual functions, risk of fall questionnaires and vision-specific quality of life questionnaire.

This project is funded by Carl Zeiss Meditec AG, led by the University of Plymouth and sponsored by University Hospitals Plymouth NHS Trust . The project also involves collaboration with the University of Glasgow and the Plymouth Marjon University.

ELIGIBILITY:
Inclusion Criteria:

* bilateral significant corneal astigmatism >1.0D
* on waiting list for bilateral cataract surgery in NHS

Exclusion Criteria:

* pre-existing eye pathology which may be aggravated by intraocular implant
* previous intraocular/ corneal surgery
* History of uveitis, glaucoma, proliferative diabetic retinopathy or IDDM, pseudoexfoliation, macular degeneration that may affect potential best corrected visual acuity of 20/40 or better
* Micropthalmia
* corneal decompensation or endothelial insufficiency
* pars planitis
* high myopia
* participants using a systematic medication that is known to cause ocular side effects
* participated in a concurrent clinical trial or have participated in an opthalmology clinical trial within the last 30 days
* unable or not willing to cooperate for the follow up period
* pregnant women
* unable to give informed consent
* unable to walk with or without walking aids independently for at least 20m
* unable to walk up/down stairs independently using aids or handrail

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Jerk from the centre of mass Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Assessed during functional activities using accelerometers
Jerk from the centre of mass Visit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  Assessed during functional activities using accelerometers
Jerk from the centre of mass Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Assessed during functional activities using accelerometers

SECONDARY OUTCOMES:
Unaided vision Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Unaided vision measured on a LogMAR acuity chart
Unaided visionVisit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  Unaided vision measured on a LogMAR acuity chart
Unaided vision Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Unaided vision measured on a LogMAR acuity chart
Visual acuity Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Aided vision measured on a LogMAR acuity chart
Visual acuity Visit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  Aided vision measured on a LogMAR acuity chart
Visual acuity Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Aided vision measured on a LogMAR acuity chart
Mean spherical refraction Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Mean spherical refraction assessed through subjective refraction
Mean spherical refraction Visit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  Mean spherical refraction assessed through subjective refraction
Mean spherical refraction Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Mean spherical refraction assessed through subjective refraction
Astigmatic power J0 Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  J0 assessed through subjective refraction and expressed in vector form
Astigmatic power J0 Visit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  J0 assessed through subjective refraction and expressed in vector form
Astigmatic power J0 Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  J0 assessed through subjective refraction and expressed in vector form
Astigmatic power J45 Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  J45 assessed through subjective refraction and expressed in vector form
Astigmatic power J45 Visit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  J45 assessed through subjective refraction and expressed in vector form
Astigmatic power J45 Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  J45 assessed through subjective refraction and expressed in vector form
Contrast sensitivity Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Contrast sensitivity measured in log units
Contrast sensitivity Visit 2 | First reassessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  Contrast sensitivity measured in log units
Contrast sensitivity Visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Contrast sensitivity measured in log units
Rotation of IOL at visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Rotation of IOL relative to operation
Rotation of IOL at visit 2 | First assessment will be carried out at study visit 2 around 3-6 months after the first cataract IOL replacement surgery
  Rotation of IOL relative to operation
Rotation of IOL at visit 3 | Final reassessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Rotation of IOL relative to Operation
Tilt of IOL at Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Tilt of IOL assessed using image analysis
Tilt of IOL at Visit 2 | assessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Tilt of IOL assessed using image analysis
Tilt of IOL at Visit 3 | assessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Tilt of IOL assessed using image analysis
Centration of IOL at Visit 1 | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Centration of IOL assessed using image analysis
Centration of IOL at Visit 2 | assessment at study visit 2 around 3-6 months after the first eye cataract IOL replacement surgery
  Centration of IOL assessed using image analysis
Centration of IOL at Visit 3 | assessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Centration of IOL assessed using image analysis
Fear of falling | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Fear of falling measured using revised fear of falling questionnaire (FFR)
Fear of falling | assessment at study visit 2 around 3-6 months after the first eye cataract IOL replacement surgery
  Fear of falling measured using revised fear of falling questionnaire (FFR)
Fear of falling | assessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Fear of falling measured using revised fear of falling questionnaire (FFR)
Risk of fall | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Risk of fall in daily activities measured by Short Fall Efficacy Scale Questionnaire (Short FFS-I)
Risk of fall | assessment at study visit 2 around 3-6 months after the first eye cataract IOL replacement surgery
  Risk of fall in daily activities measured by Short Fall Efficacy Scale Questionnaire (Short FFS-I)
Risk of fall | assessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Risk of fall in daily activities measured by Short Fall Efficacy Scale Questionnaire (Short FFS-I)
Cataract related quality of life | Baseline assessment will be carried out at study visit 1 before the cataract surgery
  Using Catract patient reported outcome measure CAT-PROM5 questionnaire
Cataract related quality of life | assessment at study visit 2 around 3-6 months after the first eye cataract IOL replacement surgery
  Using Catract patient reported outcome measure CAT-PROM5 questionnaire
Cataract related quality of life | assessment at study visit 3 around 3-6 months after the second eye cataract IOL replacement surgery
  Using Catract patient reported outcome measure CAT-PROM5 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Habib, MB ChB(Hons), Principal Investigator — Royal Eye Infirmay, University Hosptials Plymouth NHS Trust; Phillip Buckhurst, PhD, Study Chair — University of Plymouth; Catriona MacLennan, PhD, Study Director — Glasgow Caledonian Unviersity; Gary L.K. Shum, PhD, Study Director — Plymouth Marjon University; Hetal Buckhurst, PhD, Study Director — University of Plymouth
Locations (1):
- Royal Eye Infirmary, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05629078/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05629078/ICF_001.pdf